CLINICAL TRIAL: NCT02645591
Title: Neurovascular Bundle Protection With an Amnion/Chorion Membrane Allograft to Improve Postoperative Functional Recovery: A Randomized Comparison to Standard Techniques
Brief Title: Randomized AmnioFix Study During Radical Prostatectomy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-0633; NCI-2016-00342 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-12-31; First posted 2016-01-01 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Dehydrated human amnion/chorion membrane; dHACM; Robotic assisted laparoscopic radical prostatectomy; RARP; AmnioFix®; Sexual function score; Neurovascular bundle inflammation; Questionnaire; Survey
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nerve Sparing RARP + AmnioFix® (Experimental): Participants receive Nerve Sparing robotic assisted laparoscopic radical prostatectomy (RARP) plus placement of a 2x12 sheet of AmnioFix® to the neurovascular bundle.
  Interventions: Procedure: Robotic Assisted Laparoscopic Radical Prostatectomy (RARP); Biological: AmnioFix®; Behavioral: Questionnaire
- Nerve Sparing RARP (Active Comparator): Participants receive Nerve Sparing robotic assisted laparoscopic radical prostatectomy (RARP)
  Interventions: Procedure: Robotic Assisted Laparoscopic Radical Prostatectomy (RARP); Behavioral: Questionnaire

INTERVENTIONS:
Procedure: Robotic Assisted Laparoscopic Radical Prostatectomy (RARP) — Participants receive Nerve Sparing robotic assisted laparoscopic radical prostatectomy (RARP).
  Other Names: RALP
Biological: AmnioFix® — Dehydrated human amnion/chorion membrane (dHACM) wrapped around the nerve bundles at the end of Nerve Sparing robotic assisted laparoscopic radical prostatectomy (RARP) surgery.
  Other Names: Dehydrated Human Amnion/chorion Membrane; dHACM
  Arms: Nerve Sparing RARP + AmnioFix®
Behavioral: Questionnaire — Questionnaire completed about erectile function before surgery, and at 6 weeks, 3 months, 6 months, and 12 months after surgery.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to learn about the safety and the effectiveness of using AmnioFix® (dehydrated human amnion/chorion membrane, also called dHACM) to help improve the return of erectile function and bladder control in patients after robotic assisted laparoscopic radical prostatectomy (RARP).

dHACM is a section of tissue made from part of the placenta donated by a mother during a C-section. It looks like a small piece of tissue paper and is wrapped around the nerve bundles in the surgical area. The tissue may help the body's normal healing process.

DETAILED DESCRIPTION:
Study Groups:

If participant is eligible and agrees to take part in the study, they will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. Participant will have an equal chance of being in either group. This is done because no one knows if one study group is better, the same, or worse than the other group:

* If participant is in Group 1, they will have RARP with dHACM.
* If participant is in Group 2, they will have RARP alone.

Participant will not be told which group they are assigned to until they reach the end of the study. Participant will sign a separate consent form for the surgery that explains the risks.

During Surgery:

If participant is in Group 1, the dHACM will be wrapped around the nerve bundles at the end of the surgery.

For both groups, during the surgery, participant's surgeon may decide that RARP is not possible. In this case, participant will be taken off the study and dHACM will not be used.

Information will also be collected during participant's surgery, such as details about their surgery, their hospital stay, and about any side effects that they may have.

Study Visits:

Participant will visit the study doctor for their standard follow-up visits after surgery at 6 weeks, 3 months, 6 months, and 12 months. At these visits, participant will complete the same questionnaire they completed at screening.

At 24 months, participant's medical chart will be reviewed or they will be called on the phone to learn if the disease came back. If participant is called, the call should last about 5-10 minutes.

Length of Study Participation:

Patient's participation in the study will be over after the 24-month medical chart review or call.

This is an investigational study. The dHACM is commercially available for use in various types of surgeries. Its use in prostate surgery to help improve the return of erectile function and bladder control in patients after RARP is investigational.

Up to 100 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects between the ages 35-75
2. Primary diagnosis of prostate cancer selected for surgical intervention by one of the six protocol surgeons (Chapin, Davis, Matin, Pettaway, Pisters, Ward).
3. Have a willingness to comply with follow-up HRQOL (health related quality of life) surveys and PSA assessments.
4. Have ability to provide full written consent.
5. Primary diagnosis of untreated with clinically localized prostate cancer with Gleason score of 6, 7,8 or 9.
6. Planned elective radical prostatectomy with bilateral nerve sparing technique that can include high or low fascia.
7. Negative urinalysis within 30 days prior to date of surgery

Exclusion Criteria:

1. High-risk cancer planned for neoadjuvant therapy, full or partial excision of one or both neurovascular bundles.
2. Has any condition(s), which seriously compromises the subject's ability to participate in this study, sign consent, or has a known history of poor adherence with medical treatment.
3. Is unable to comply with learning and documenting penile rehabilitation, including oral 5-phosphodiesterase inhibitor use, vacuum pump therapy use, and/or injectable medications.
4. In the opinion of the PI, has a history of drug or alcohol abuse within last 12 months.
5. Is allergic to Aminoglycoside antibiotics (such as Gentamicin and/or Streptomycin).
6. Patients with a history of more than two weeks treatment with immuno-suppressants (including systemic corticosteroids), cytotoxic chemotherapy within one month prior to initial screening, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
7. Patients currently enrolled in another study. Concurrent enrollment in another study is prohibited expect for the control arm which can be used for other protocols with HRQOL endpoints with similar instruments.
8. Has had prior hormonal therapy such as Lupron or oral anti-androgens.
9. Unwilling to participate in follow-up clinical appointments at MDACC.

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Reducing Neurovascular Bundle Inflammation in Prostate Cancer Patients Undergoing Nerve Sparing Robotic Assisted Laparoscopic Radical Prostatectomy (RARP) | 3 months
  Outcome determined by a 10-point improvement in 3-month post-prostatectomy sexual function score using the Expanded Prostate Cancer Index Composite (EPIC) 26 in patients treated with the AmnioFix® graft compared to standard treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John W. Davis, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org